CLINICAL TRIAL: NCT01787357
Title: A Randomized, Double-Blind, Double-Dummy, Placebo- and Positive-Controlled, Four-Way Crossover Study Evaluating ECG Intervals in Healthy Adults Receiving a Single, Oral Dose of JNJ-28431754 at Therapeutic and Supra-Therapeutic Doses
Brief Title: A Study to Assess Electrocardiogram Results in Healthy Volunteers Receiving Canagliflozin (JNJ-28431754)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR015514; 28431754DIA1010 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: Healthy; Canagliflozin (JNJ-28431754); Pharmacokinetics; Moxifloxacin; Electrocardiogram Parameters; QT/QTc Interval; Therapeutic dose; Supra-Therapeutic dose
MeSH Terms: interventions — Canagliflozin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (ADBC) (Experimental): Each volunteer will receive Treatment A on Day 1 of Treatment Period 1, followed by Treatment D on Day 1 of Treatment Period 2, followed by Teatment B on Day 1 of Treatment Period 3, and followed by Treatment C on Day 1 of Treatment Period 4. Each treatment period will be 2 days in duration and there will be a washout period (with no medication) of 10 to 14 days between each treatment period.
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Placebo; Drug: Moxifloxacin
- Sequence 2 (BACD) (Experimental): Each volunteer will receive Treatment B on Day 1 of Treatment Period 1, followed by Treatment A on Day 1 of Treatment Period 2, followed by Treatment C on Day 1 of Treatment Period 3, and followed by Treatment D on Day 1 of Treatment Period 4. Each treatment period will be 2 days in duration and there will be a washout period (with no medication) of 10 to 14 days between each treatment period.
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Placebo; Drug: Moxifloxacin
- Sequence 3 (CBDA) (Experimental): Each volunteer will receive Treatment C on Day 1 of Treatment Period 1, followed by Treatment B on Day 1 of Treatment Period 2, followed by Treatment D on Day 1 of Treatment Period 3, and followed by Treatment A on Day 1 of Treatment Period 4. Each treatment period will be 2 days in duration and there will be a washout period (with no medication) of 10 to 14 days between each treatment period.
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Placebo; Drug: Moxifloxacin
- Sequence 4 (DCAB) (Experimental): Each volunteer will receive Treatment D on Day 1 of Treatment Period 1, followed by Treatment C on Day 1 of Treatment Period 2, followed by Treatment A on Day 1 of Treatment Period 3, and followed by Treatment B on Day 1 of Treatment Period 4. Each treatment period will be 2 days in duration and there will be a washout period (with no medication) of 10 to 14 days between each treatment period.
  Interventions: Drug: Canagliflozin (JNJ-28431754); Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Canagliflozin (JNJ-28431754) — One 300 mg dose of canagliflozin (JNJ-28431754) (comprising one 100 mg over-encapsulated tablet and one 200 mg over-encapsulated tablet) taken orally (by mouth) on Day 1 of Treatment A. One 1,200 mg dose of canagliflozin (comprising six 200 mg over-encapsulated tablets) taken orally on Day 1 of Treatment B.
  Other Names: JNJ-28431754
Drug: Placebo — Four over-encapsulated matching placebo tablets taken orally (by mouth) on Day 1 of Treatment A. Six over-encapsulated matching placebo tablets taken orally on Day 1 of Treatment C. Five encapsulated matching placebo tablets taken orally on Day 1 of Treatment D.
Drug: Moxifloxacin — One 400 mg over-encapsulated tablet of moxifloxacin taken orally (by mouth) on Day 1 of Treatment D.

SUMMARY:
The purpose of this study is to assess the effect of canagliflozin (JNJ-28431754) on electrocardiogram results (recordings of the electrical activity of the heart) in healthy volunteers after a single therapeutic dose (300 mg) and a single supra-therapeutic dose (4 times higher [1,200 mg] than the anticipated therapeutic dose of 300 mg). The safety and tolerability of canagliflozin will also be assessed.

DETAILED DESCRIPTION:
This study will be a randomized (the treatment is assigned by chance), single-center, double-blind (neither investigator nor volunteer knows the identity of the assigned treatment), double-dummy (a technique for retaining the blinded nature of the study when the treatments do not look identical), placebo-controlled (one of the treatments is inactive), positive-controlled (one of the treatments has a known potential effect on electrocardiogram results), four-way cross-over study (all volunteers will receive each of the 4 treatments but in a different order) to assess the effect of canagliflozin (a drug currently being investigated for the treatment of type 2 diabetes mellitus) on electrocardiogram results in healthy volunteers. The study will consist of 3 phases: a screening phase, a double-blind treatment phase, and an end-of study (or follow-up) phase. Volunteers will be assigned to 1 of 4 treatment sequence groups (ADBC, DABC, BCDA, or CDAB). The treatment sequence will be decided by randomization. Treatment A will be a single dose of 300 mg of canagliflozin. Treatment B will be a single dose of 1,200 mg of canagliflozin. Treatment C will be a single dose of placebo (inactive medication). Treatment D will be a single dose of 400 mg of moxifloxacin (an antibiotic with known potential to affect electrocardiogram results). Each treatment will be given during a treatment period of 2 days duration; each treatment period will be separated by a washout period (when no medication is given) of 10 to 14 days. Each volunteer will participate in the study for approximately 61 days.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must have a body mass index (BMI = weight in kg/height in m2) between 18 and 35 kg/m2 (inclusive) and body weight not less than 50 kg
* Volunteers must have an average of triplicate 12-lead electrocardiogram (ECG) recordings, taken with a maximum of 2 minutes between recordings, consistent with normal cardiac conduction and function, as specified by the protocol
* Volunteers must be non-smokers

Exclusion Criteria:

* History of or currently active illness considered to be clinically significant by the Investigator or any other illness that the Investigator considers should exclude the patient from the study or that could interfere with the interpretation of the study results
* History of additional risk factors for the presence of a family history of Short QT Syndrome, Long QT Syndrome, sudden unexplained death at a young age (<=40 years), drowning or sudden infant death syndrome in a first degree relative (ie, biological parent, sibling, or child)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTc intervals | Day 1 (Predose) up to Day 2
  QT intervals (assessment of the electrical activity of the heart) will be measured from 12-lead electrocardiogram (ECG) readings and will be corrected for heart rate. The corrected QT intervals (QTc) obtained following single doses of 300 mg canagliflozin (JNJ-28431754), 1,200 mg canagliflozin, and 400 mg moxifloxacin, will be compared with QTc intervals obtained following dosing with placebo.

SECONDARY OUTCOMES:
Number of volunteers with adverse events | Up to 61 days
  Adverse events will be used as a measure of safety and tolerability.
Plasma concentrations of canagliflozin (JNJ-28431754) | Up to Day 2
  Plasma concentrations of canagliflozin (JNJ-28431754), following the administration of a single 300 mg dose and a single 1,200 mg dose, will be used to determine pharmacokinetic parameters for canagliflozin (measurements describing how the body affects the drug).
QRS intervals obtained from 12-lead electrocardiogram (ECG) readings | Up to Day 2
  QRS intervals will be obtained from 12-lead electrocardiogram (ECG) readings following a single 300 mg dose and a single 1,200 mg dose of canagliflozin (JNJ-28431754).
PR intervals obtained from 12-lead electrocardiogram (ECG) readings | Up to Day 2
  PR intervals will be obtained from 12-lead electrocardiogram (ECG) readings following a single 300 mg dose and a single 1,200 mg dose of canagliflozin (JNJ-28431754).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Tempe, Arizona, United States

REFERENCES:
- See also: A Randomized, Double-Blind, Double-Dummy, Placebo- and Positive-Controlled, Four-Way Crossover Study Evaluating Electrocardiogram Intervals in Healthy Adults Receiving a Single, Oral Dose of JNJ-28431754 at Therapeutic and Supra-Therapeutic Doses — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=2261&filename=CR015514_CSR.pdf